CLINICAL TRIAL: NCT07283172
Title: The Effect of Virtual Reality on Pain and Anxiety During Chest Tube Removal in Patients With Cardiac Surgery
Brief Title: The Effect of Virtual Reality
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Collaborators: Giresun University Funding for Scientific Research Project (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: BAEK-492
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: The Effects of Virtual Reality on Pain and Anxiety Levels During Chest Tube Removal
Keywords: Cardiac Surgery; Chest Tube; Virtual Reality; Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Control Group
- Virtual Reality Group (Experimental): Virtual Reality Group
  Interventions: Other: Virtual Reality

INTERVENTIONS:
Other: Virtual Reality — Fifteen minutes before the chest tube removal procedure begins, patients' pain intensity will be measured using the "Visual Analog Scale (VAS)" and their anxiety level will be measured using the "State Anxiety Inventory" (1st MEASUREMENT). The researcher will provide each patient in the intervention group with detailed information about the virtual reality application, how to use the headset, what to do, the video content, and the procedure to be performed before the virtual reality application. Five minutes before the procedure, the virtual reality headset will be put on and the video will be shown. During the virtual reality application, all chest tubes will be removed by the physician. Immediately after the chest tube is removed, the intensity of pain felt by the patient during tube removal will be measured again using the VAS (2nd MEASUREMENT). Twenty minutes after the chest tube is removed, the patient's pain intensity will be measured again using the VAS, and their anxiety level
  Arms: Virtual Reality Group

SUMMARY:
Chest tubes are routinely required during cardiothoracic procedures in open-heart surgeries. Postoperatively, these tubes are typically removed within 24-48 hours, and the removal process often causes patients to experience significant pain and discomfort due to the force applied. Among non-pharmacological strategies for managing procedural pain, distraction techniques are commonly used to divert patients' attention away from painful stimuli. In this context, the use of virtual reality (VR) headsets has recently emerged as an innovative method for pain management, effectively redirecting attention during invasive interventions.

The aim of this study is to evaluate the effects of virtual reality on pain and anxiety levels during chest tube removal. This research is designed as a randomized controlled experimental trial. The study population will consist of patients undergoing open-heart surgery at the Cardiovascular Surgery Clinic of Giresun Training and Research Hospital. A total of 60 patients who meet the inclusion criteria and are representative of the study population will be recruited. Data will be collected using a Patient Identification Form developed by the researchers to assess sociodemographic characteristics, the Visual Analog Scale (VAS), and the State Anxiety Inventory. Participants will be randomly assigned to either the experimental or control group. Patients in the control group will receive routine care without additional intervention. In the experimental group, patients will be thoroughly informed about the VR procedure, including instructions on how to use the headset, details of the video content, and an explanation of the upcoming intervention. Five minutes before chest tube removal, the VR headset will be placed on the patient, and a video will be shown. The physician will then remove the chest tube(s) while the patient is engaged in the VR session. Pain intensity will be assessed at three time points: before chest tube removal, immediately after the procedure, and 20 minutes post-procedure. Anxiety levels will be evaluated twice: before the procedure and 20 minutes afterward. Data will be analyzed using SPSS version 22.0. Descriptive statistics, chi-square tests, and independent t-tests will be used for group comparisons, while repeated measures analysis of variance (R-ANOVA) will be employed for repeated measures.

DETAILED DESCRIPTION:
The prevalence of coronary artery disease is increasing, and during open-heart surgery, a chest tube is required and used in cardiopulmonary bypass procedures. A chest tube is applied to drain air and fluid accumulated in the pleural space after open heart surgery, reduce the size of the pleural space, return the pleural space pressure to normal and restore negative pressure, ensure normal ventilation in the lungs, prevent mediastinal shift, and prevent the return of air and fluid accumulated in the drainage system. Chest tubes can be placed behind the pectoralis major muscle from the area where the 3rd and 5th intercostal spaces intersect with the midaxillary line, either bilaterally or unilaterally depending on the surgical procedure and the disease. Postoperatively, chest tubes are usually removed 24-48 hours later when the fluid becomes serous or when the amount of fluid collected in 24 hours is less than 150 ml. Since chest tubes adhere to the endothelium after being placed in the pleural space, the force applied during removal causes the patient to experience significant pain and discomfort.

Nurses play the most significant role in pain management as they are the healthcare professionals most involved in patient care and spend the most time with patients. Managing the procedural pain experienced during chest tube removal increases the patient's comfort level. For pain management to be effective, nurses must possess the correct knowledge, behavior, attitude, assessment, and decision-making skills. Both pharmacological and nonpharmacological methods are used in pain management. Due to its rapid effect and ease of application, analgesia is the most preferred method for pain relief. However, non-pharmacological methods reduce the use of analgesics and increase patient comfort by reducing pain. These methods offer advantages such as no side effects like analgesic drugs, no economic burden, and ease of application.

The distraction technique, which holds an important place among non-pharmacological methods, aims to reduce pain perception by preventing the patient from focusing on the painful stimulus. In this context, virtual reality applications stand out as a powerful distraction method. Through virtual reality, the patient's attention is directed away from the pain and the painful treatment process and toward alternative visual and auditory stimuli; thus, the sensation of pain is alleviated, and the goal is to reduce pain-related fear and anxiety. Virtual reality is defined as a dynamic simulation environment that provides an individual with a sense of reality through a computer-based interface that appeals to visual, auditory, and sometimes tactile senses, offering the possibility of interactive engagement.

Various studies have been conducted in the literature on procedural pain and anxiety experienced during chest tube removal. However, it is noteworthy that studies using technology-based innovative applications, such as virtual reality, and evaluating the effects of these applications are limited. The primary objective of this study is to demonstrate the integration and applicability of virtual reality technology, which makes significant contributions to healthcare services today, with nursing care processes. The study aims to introduce a new approach to patient care and enhance patient comfort by examining the effects of virtual reality applications on pain and anxiety during chest tube removal.

The findings obtained from the research will shed light on the feasibility of using virtual reality applications as an effective support tool for pain and anxiety management in clinical settings. This will contribute to minimizing the negative experiences patients encounter during invasive procedures and creating a more positive patient experience during the treatment process. Furthermore, the study will significantly contribute to raising awareness of digital health applications and filling existing scientific gaps in this field by promoting the integration of technology with nursing practices. As a result, this research will enhance patient comfort and safety while developing a sustainable, innovative, and contemporary approach to improving the quality of healthcare services.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Undergone open heart surgery and have a chest tube,
* Able to communicate verbally,
* Have not previously received any psychiatric diagnosis or treatment and are not taking psychiatric medication,
* Hemodynamic status is stable,
* Patients who agree to participate in the study will be included.

Exclusion Criteria:

* Patients who used analgesic medication immediately before the chest tube removal procedure,
* Patients with a history of chronic pain who routinely use analgesic medication,
* Patients who wear prescription glasses and have vision problems will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Participants' pain intensity (VAS) will be assessed three times: before chest tube removal, immediately after the procedure, and 20 minutes after the procedure.
  Visual Analog Scale (VAS) will be used to assess procedural pain. The VAS, which has undergone psychometric evaluation, is used to assess acute pain intensity in various patient populations, particularly to evaluate the effectiveness of treatment/intervention. In addition, many authors recommend using the VAS to measure the intensity of acute pain experienced during chest tube removal because it is easier and more understandable. The VAS is a 10 cm long scale that can be used horizontally or vertically, starting with "no pain" and ending with "unbearable pain."

SECONDARY OUTCOMES:
State Anxiety Inventory | Patients' anxiety levels will be assessed before the chest tube removal procedure and 20 minutes after the procedure.
  This is a 4-point Likert-type inventory consisting of 20 items that aims to determine how an individual feels at a given moment and under specific conditions. In the State Anxiety Inventory, the individual is asked to assess how they feel "right now" and to select one of the following statements based on the intensity of the feelings or behaviors expressed in the items: (1) "not at all," (2) "a little," (3) "a lot," and (4) "completely." A score of 4 is given for selecting "completely," and a score of 1 is given for selecting "not at all." A high score indicates a high level of anxiety, while a low score indicates a low level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Yeşim Yaman Aktaş, Professor, Principal Investigator — Giresun University
Locations (1):
- Giresun University Health Sciences Faculty, Giresun, Piraziz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kok AY, Eyiler E. Effectiveness of breathing relaxation exercises on pain due to chest tube removal: a systematic review-meta-analysis. J Cardiothorac Surg. 2025 Jul 2;20(1):281. doi: 10.1186/s13019-025-03444-4. PMID 40604937
- [Result] Tsai CS, Tung HH, Fang CJ, Chen CT. Effectiveness of non-pharmacological interventions for pain reduction following chest tube removal: A systematic review and network meta-analysis. Intensive Crit Care Nurs. 2025 Apr;87:103909. doi: 10.1016/j.iccn.2024.103909. Epub 2024 Nov 29. PMID 39615184
- [Result] Demir Y, Khorshid L. The effect of cold application in combination with standard analgesic administration on pain and anxiety during chest tube removal: a single-blinded, randomized, double-controlled study. Pain Manag Nurs. 2010 Sep;11(3):186-96. doi: 10.1016/j.pmn.2009.09.002. Epub 2010 May 31. PMID 20728068
- [Result] Andreasen JJ, Sorensen GV, Abrahamsen ER, Hansen-Nord E, Bundgaard K, Bendtsen MD, Troelsen P. Early chest tube removal following cardiac surgery is associated with pleural and/or pericardial effusions requiring invasive treatment. Eur J Cardiothorac Surg. 2016 Jan;49(1):288-92. doi: 10.1093/ejcts/ezv005. Epub 2015 Feb 7. PMID 25661079